CLINICAL TRIAL: NCT01819012
Title: Effect of Isoflurane on Tissue Doppler Imaging of Mitral Annulus During Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KUH1160052
Record Dates: First submitted 2013-03-22; First posted 2013-03-27 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Valvular Heart Disease; Ischemic Heart Disease
Keywords: Isoflurane; mitral valve annular velocity; tissue Doppler imaging; Monitoring; echocardiography
MeSH Terms: conditions — Heart Valve Diseases; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Isoflurane 1.0 MAC (Experimental): 10 min-inhalation of each concentration of isoflurane, 1.0 MAC
  Interventions: Drug: Isoflurane 1.0 MAC
- Isoflurane 1.5 MAC (Experimental): 10 min-inhalation of each concentration of isoflurane, 1.5 MAC
  Interventions: Drug: Isoflurane 1.5 MAC
- Isoflurane 2.0 MAC (Experimental): 10 min-inhalation of each concentration of isoflurane, 2.0 MAC
  Interventions: Drug: Isoflurane 2.0 MAC

INTERVENTIONS:
Drug: Isoflurane 1.0 MAC — 10 min-inhalation of each concentration of isoflurane, 1.0 MAC
  Arms: Isoflurane 1.0 MAC
Drug: Isoflurane 1.5 MAC — 10 min-inhalation of each concentration of isoflurane, 1.5 MAC
  Arms: Isoflurane 1.5 MAC
Drug: Isoflurane 2.0 MAC — 10 min-inhalation of each concentration of isoflurane, 2.0 MAC
  Arms: Isoflurane 2.0 MAC

SUMMARY:
The purpose of this study is to determine Isoflurane's dose-dependent effect on left ventricular (LV) systolic function in cardiac surgery. The change of tissue Doppler imaging (TDI) of lateral mitral valve annular systolic velocity at three different isoflurane concentrations would be analyzed by using intraoperative transesophageal echocardiography (TEE) in cardiac surgery patients.

DETAILED DESCRIPTION:
Isoflurane is widely used in cardiac surgery patients due to its beneficial effects, but many studies have shown that isoflurane reduces myocardial contractility in a dose-dependent manner, and compromises left ventricular (LV) function.

Tissue Doppler imaging (TDI) of mitral annular velocity during the cardiac cycle has been introduced as a reliable method for analysis of systolic and diastolic LV long-axis function. Efficacy of systolic and diastolic TDI profiles, including systole (S'), early early relaxation (E')and atrial contraction (A') have been suggested to be useful in predicting the impact of isoflurane on LV systolic and diastolic function.

The investigators hypothesized that isoflurane, even at a clinical dosage, would affects intraoperative LV systolic function in a dose-dependent manner and thus produce significant changes int the TDI profiles of systolic mitral annular velocity (S').

So the investigators planned to study the changes in S' of lateral mitral annulus at the clinical isoflurane dosage during remifentanil based anesthesia for cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cardiac surgery

Exclusion Criteria:

* low ejection fraction < 50% in preoperative transthoracic echocardiography
* atrial fibrillation
* pacemaker
* pericardial and infiltrative myocardial disease
* mitral annular calcification, surgical rings, prosthetic mitral valves
* lateral left ventricular regional wall motion abnormality
* esophageal spasm, stricture, laceration, perforation, and diverticulum diaphragmatic hernia
* history of extensive radiation to mediastinum
* upper gastrointestinal bleeding

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Peak mitral annular velocity during systole(S') | after 10 min exposure to isoflurane 1.0 MAC, 1.5 MAC and 2.0 MAC
  By using pulsed Doppler with the sample volume positioned at the lateral mitral valve (MV)ring in the midesophageal 4-chamber view, S' would be determined just after the 10 min-exposure to each concentration of isoflurane, 1.0 MAC, 1.5 MAC and 2.0 MAC (T1, T2 and T3, respectively)

SECONDARY OUTCOMES:
ejection fraction(EF) | after 10 min exposure to isoflurane 1.0 MAC, 1.5 MAC and 2.0 MAC
  By using modified Simpson technique in the midesophageal 4-chamber view, EF would be determined just after the 10 min-exposure to each concentration of isoflurane 1.0 MAC, 1.5 MAC and 2.0 MAC
bispectral index(BIS) | after 10 min exposure to isoflurane 1.0 MAC, 1.5 MAC and 2.0 MAC
  BIS would be determined just after the 10 min-exposure to each concentration of isoflurane 1.0 MAC, 1.5 MAC and 2.0 MAC
peak velocity of mitral inflow during early relaxation(E) | after 10 min exposure to isoflurane 1.0 MAC, 1.5 MAC and 2.0 MAC
  By using pulsed Doppler with the sample volume positioned at the IMV opening in the midesophageal 4-chamber view, E' would be determined just after the 10 min-exposure to each concentration of isoflurane, 1.0 MAC, 1.5 MAC and 2.0 MAC(T1, T2 and T3, respectively)
peak velocity of mitral inflow during atrial contraction(A) | after 10 min exposure to isoflurane 1.0 MAC, 1.5 MAC and 2.0 MAC
  By using pulsed Doppler with the sample volume positioned at the tip of MV opening in the midesophageal 4-chamber view, "A" would be determined just after the 10 min-exposure to each concentration of isoflurane, 1.0 MAC, 1.5 MAC and 2.0 MAC(T1, T2 and T3, respectively)
Peak mitral annular velocity during early diastole(E') | after 10 min exposure to isoflurane 1.0 MAC, 1.5 MAC and 2.0 MAC
  By using pulsed Doppler with the sample volume positioned at the lateral MV ring
Peak mitral annular velocity during atrial contraction(A') | after 10 min exposure to isoflurane 1.0 MAC, 1.5 MAC and 2.0 MAC
  By using pulsed Doppler with the sample volume positioned at the lateral MV ring

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Yop Kim, MD, PhD, Principal Investigator — Konkuk University
Locations (1):
- Konkuk University Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JD, Son I, Kwon WK, Sung TY, Sidik H, Kim K, Kang H, Bang J, Yeo GE, Lee DK, Kim TY. Isoflurane's Effect on Intraoperative Systolic Left Ventricular Performance in Cardiac Valve Surgery Patients. J Korean Med Sci. 2018 Jan 22;33(4):e28. doi: 10.3346/jkms.2018.33.e28. PMID 29318795